CLINICAL TRIAL: NCT01218217
Title: A Phase 2A Trial to Evaluate the Extended Early Bactericidal Activity, Safety, Tolerability, and Pharmacokinetics of SQ109 in Adult Subjects With Newly Diagnosed, Uncomplicated, Smear-Positive, Pulmonary Tuberculosis
Brief Title: Early Bactericidal Activity (EBA) of SQ109 in Adult Subjects With Pulmonary TB
Acronym: SQ109EBA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michael Hoelscher (Other)
Collaborators: Sequella, Inc. (Industry); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); German Federal Ministry of Education and Research (Other Government); Quintiles, Inc. (Industry); CMed Technologies Inc. (Industry); PathCare (Unknown); Parexel (Industry)
Responsible Party: Sponsor-Investigator, Michael Hoelscher, Professor, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LMU-IMPH-SQ109-01
Record Dates: First submitted 2010-10-08; First posted 2010-10-11 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Tuberculosis, Pulmonary
Keywords: TB; Tuberculosis; EBA; Pulmonary; Early Bactericidal Activity
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis | interventions — Rifampin

ARMS (6):
- SQ109 75 mg (Experimental): 75 mg SQ109 monotherapy daily
  Interventions: Drug: SQ109
- SQ109 150 mg (Experimental): 150 mg SQ109 daily
  Interventions: Drug: SQ109
- SQ109 300 mg (Experimental): 300 mg SQ109 daily
  Interventions: Drug: SQ109
- SQ109 150 mg + RIF (Experimental): 150 mg SQ109 + RIF standard dose daily
  Interventions: Drug: SQ109; Drug: Rifampicin
- SQ109 300 mg + RIF (Experimental): 300 mg SQ109 + RIF standard dose daily
  Interventions: Drug: SQ109; Drug: Rifampicin
- RIF Mono (Active Comparator): Standard dose Rifampicin monotherapy daily
  Interventions: Drug: Rifampicin

INTERVENTIONS:
Drug: SQ109 — SQ109 150 mg tablet
  Arms: SQ109 150 mg; SQ109 150 mg + RIF; SQ109 300 mg; SQ109 300 mg + RIF; SQ109 75 mg
Drug: Rifampicin — Rifampicin 150 mg capsules
  Arms: RIF Mono; SQ109 150 mg + RIF; SQ109 300 mg + RIF

SUMMARY:
SQ109 was developed with the aim of shortening TB treatment and providing new drugs for resistant TB. The drug has demonstrated efficacy in toxicology studies and an acceptable safety profile in first-in-man studies. The objective of this study is to evaluate the extended early bactericidal activity (EBA), safety, tolerability, and pharmacokinetics of several doses of SQ109 with or without Rifampicin (RIF) for 14 days in adults with newly diagnosed, uncomplicated, smear positive, pulmonary TB.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed written informed consent for study participation, including HIV testing (if HIV serostatus is not known or the last documented negative is more than four weeks prior to enrolment).
2. Be eighteen (18) to 64 (inclusive) years of age.
3. Have a body weight (in light clothing and with no shoes) between 40 and 90 kg, inclusive.
4. Have newly diagnosed, previously untreated, uncomplicated, sputum smear-positive, pulmonary TB.
5. Have a chest X-ray which, in the opinion of the Investigator, is compatible with TB.
6. Is sputum positive on direct microscopy for acid-fast bacilli (at least 1+ on the IUATLD/WHO scale (Appendix 3).
7. Is able to produce an adequate spot sputum sample, indicating an overnight sputum volume of at least 10 mL.
8. Female patients of childbearing potential must have a negative serum pregnancy test, and consent to practice two effective methods of birth control when not abstaining from sexual intercourse, unless she and her partner(s) are surgically sterile or she is post-menopausal with no menses for the last 12 months. Preferably, contraceptive measures should be continued until completion of TB treatment, but at least until one month after last dose of IMP, unless she and her partner(s) are sterile (that is, women who have had a bilateral oophorectomy or hysterectomy or have been postmenopausal for at least 12 consecutive months).

   Two of the following methods may be used, but only one may be hormonal: tubal ligation, vaginal diaphragm, intrauterine device, condom, oral contraceptives, contraceptive implant, combined hormonal patch, combined injectable contraceptive or depot-medroxyprogesterone acetate, partner(s) has had a vasectomy.
9. Male participants must agree to use an adequate method of contraception when not abstaining from sexual intercourse throughout participation in the trial and for 12 weeks after last dose, unless he has had bilateral orchidectomy.
10. A Karnofsky score of at least 60 (requires occasional assistance but is able to care for most of his/her needs, see Appendix 5)

Exclusion Criteria:

1. Poor general condition where any delay in treatment cannot be tolerated per discretion of Investigator.
2. Treatment with any drug active against MTB within the 3 months prior to Visit 1 (this includes, but is not limited to INH, EMB, RIF, PZA, amikacin, cycloserine, rifabutin, streptomycin, kanamycin, para-aminosalicylic acid, rifapentine, thioacetazone, capreomycin, fluoroquinolone, thioamides, metronidazole).
3. Sputum isolate is resistant to RIF as detected by rapid assay from native sputum
4. A history of allergy to the IMP or related substances.
5. Clinically significant evidence of extrathoracic TB (miliary TB, abdominal TB, urogenital TB, osteoarthritic TB, TB meningitis), as judged by the investigator.
6. A history of previous TB.
7. Evidence of serious lung conditions other than TB or uncontrolled obstructive bronchial disease.
8. Laboratory parameters done at, or within 14 days prior to, screening:

   * Serum amino aspartate transferase (AST) and/or serum alanine aminotransferase (ALT) activity >3 times the upper limit of normal
   * Serum total bilirubin level >2.5 times the upper limit of normal
   * Serum creatinine level >2 times the upper limit of normal
   * Complete blood count with hemoglobin level <7.0 g/dL
   * Platelet count <50,000/mm3
   * Serum potassium <3.5 meq/L
9. History, presence, or evidence of a neuropathy or epilepsy.
10. Clinically relevant change s in the ECG such as atrioventricular (AV) block, prolongation of the QRS complex over 120 milliseconds, or of either the QTcF or QTcB interval over 450 milliseconds on the screening ECG.
11. A history of, or current clinically relevant cardiovascular disorder such as myocardial infarction, heart failure, coronary heart disease, hypertension, arrhythmia, or tachyarrhythmia. Family history of sudden death of unknown or cardiac-related cause, or of prolonged QTc interval. Concomitant use of any drug known to prolong QTc interval (including amiodarone, bepridil chloroquine, chlorpromazine, cisapride, cisapride, clarithromycin, disopyramide dofetilide, domperidone, droperidol, erythromycin, halofantrine, haloperidol, ibutilide, levomethadyl, lumefantrine, mesoridazine, methadone, pentamidine, pimozide, procainamide, quinidine, sotalol, sparfloxacin, terfenadine, thioridazine).
12. Diabetics using insulin.
13. Evidence of clinically significant metabolic, gastrointestinal, neurological, psychiatric or endocrine diseases, malignancy, or other abnormalities (other than the indication being studied).
14. Any disease or condition in which the use of the standard TB drugs or any of their components is contraindicated, including but not limited to allergy to any TB drug, their components or to the IMPs.
15. Any disease or condition in which any of the medicinal products listed in the section pertaining to prohibited medication (see 4.10.4) is used.
16. Known or suspected, current or history of within the past 2 years, alcohol or drug abuse, that is, in the opinion of the investigator, sufficient to compromise the safety or cooperation of the patient. Opiates prescribed for cough relief are not counted as drug abuse.
17. Prior administration of SQ109.
18. Is pregnant, breast-feeding, or planning to conceive or father a child within one month of cessation of treatment.
19. Use of any drugs or substances within 30 days prior to dosing known to be strong inhibitors or inducers of cytochrome P450 enzymes (including xenobiotics, quinidine, tyramine, ketoconazole, testosterone, quinine, gestodene, metyrapone, phenelzine, doxorubicin, troleandomycin, cyclobenzaprine, erythromycin, cocaine, furafylline, cimetidine, dextromethorphan). Exceptions may be made for subjects that have received 3 days or less of one of these drugs or substances, if there has been a wash-out period equivalent to at least 5 half-lives of that drug or substance.
20. Use of any therapeutic agents within 30 days prior to dosing known to alter any major organ function (e.g., barbiturates, opiates, phenothiazines, cimetidine).
21. Use of systemic glucocorticoids within three months prior to dosing.
22. HIV infection with helper/inducer T lymphocyte (CD4 cell) count of 250 10-6/L.
23. Receiving antiretroviral therapy (ART).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2010-11; Primary Completion 2011-09 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
The extended early bactericidal activity (EBA)of daily 75 mg, 150 mg, and 300 mg SQ109, and of daily 150 mg or 300 mg SQ109 with daily RIF standard dose in adults with newly diagnosed, uncomplicated, smear positive, pulmonary TB. | Daily during first two weeks

SECONDARY OUTCOMES:
The standard EBA (EBA 0-2) of each treatment group, as determined by the rate of change of log Colony Forming Units (logCFU) in sputum over the period Day 0-2 (linear, bi-linear or non-linear regression of logCFU over time). | Day 0 - Day 2
Extended EBA (EBA 2-14) of each treatment group, as determined by the rate of change of logCFU in sputum over the periods Day 2-14 (linear, bi-linear or non-linear regression of logCFU over time). | Days 2-14
The change in time to positivity (TTP) in the Mycobacterium Growth Indicator Tube (Bactec MGIT 960 system). | Days 0-14
Pharmacokinetics | Days 1,2,7,8,14,15
Proportion of subjects with serious adverse events and proportion of subjects who discontinue due to an adverse event in each experimental arm. | Entire study period
  These will be presented as descriptive analyses, and no inferential tests will be carried out.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hoelscher, MD, Study Chair — Klinikum of the University of Munich; Andreas Diacon, MD, Principal Investigator — Task Applied Sciences; Rodney Dawson, MD, Principal Investigator — University of Cape Town
Locations (2):
- South Africa (2):
  - TASK Applied Sciences, Cape Town
  - University of Cape Town, Cape Town